CLINICAL TRIAL: NCT03506386
Title: Multiple Myeloma Profile in Brazil: A Retrospective Observational Analysis
Brief Title: Multiple Myeloma (MM) Profile in Brazil: A Retrospective Observational Analysis
Acronym: MMyBRave
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: NDMM-5004
Record Dates: First submitted 2018-04-19; First posted 2018-04-24 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Multiple Myeloma
Keywords: Real World Evidence , Multiple Myeloma Profile, Brazil
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Myeloma Participants: Participants with multiple myeloma (MM) were observed retrospectively since the diagnosis up to death or lost to follow-up within the eligibility window of time (between January 1, 2008 and December 31, 2016), in this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As it was an observational study, no intervention was administered.

SUMMARY:
The purpose of this study is to present a descriptive analysis of demographic and clinical characteristics of the participants, as well as of the treatment patterns for multiple myeloma (MM) in Brazil.

DETAILED DESCRIPTION:
Participants with a diagnosis of MM will be observed in this retrospective study. Data collected for the study will include identification, demographic, baseline data on MM, additional baseline laboratory, initial treatment for MM, subsequent treatment for MM, and outcome.

The study will enroll approximately 1000 participants.

This multi-center trial will be conducted in five geographic regions of Brazil. For each participant, data collection will comprise the longest possible period of time since the diagnosis of MM (within the eligibility window of time, between January 1, 2008 and December 31, 2016) and the cut-off date for data collection (December 31, 2016), unless a participant has died or been lost to follow-up before that. The study is planned to last for approximately 24 months since its initiation (initiation defined as the initiation visit for the first site).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent, for participants who are alive and not lost to follow-up (for participants already deceased or lost follow up, informed consent should have been waived by the corresponding ethics review board [ERB]).
2. Documented diagnosis of MM by the responsible physician between January 1, 2008, and December 31, 2016.
3. Absence of any plasma-cell disorder other than MM.
4. Absence of any immunoglobulin-related disorder other than MM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each participant should be included in the study only once. For study sites with a system that allows identification of participants with MM electronically, for example using International Classification of Diseases, 10th revision (ICD-10), this will be the preferred method of participant screening for eligibility. For study sites without such capabilities, participant screening will rely on manual selection of institutional charts or other means. In these cases, every effort should be made to identify every possible eligible participant.
Sampling Method: Non-Probability Sample
Enrollment: 943 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Science, Study Director — Takeda
Locations (17):
- Brazil (17):
  - Centro de Hematologia e Oncologia (CEHON), Salvador, Estado de Bahia
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Hospital das Clinicas da UFG, Goiânia, Goiás
  - Hospital das Clinicas da UFMG, Belo Horizonte, Minas Gerais
  - Fundacao IMEPEN, Juiz de Fora, Minas Gerais
  - Clinica de Tratamento e Pesquisa em Hematologia LTDA., Cuiabá, Mount
  - Hospital das Clinicas da UFPR, Curitiba, Paraná
  - CIONC - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas (CEPON), Florianópolis, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital do Servidor Publico de SP, São Paulo, São Paulo
  - Clinica Sao Germano, São Paulo, São Paulo
  - Hospital das Clinicas da FMUSP, São Paulo, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 17 investigative sites in Brazil from 9 August 2018 to 27 January 2020.
Pre-assignment Details: Participants with a diagnosis of Multiple Myeloma (MM) were observed to collect data retrospectively between eligibility window: 1 January 2008 to 31 December 2016, in this study.
Groups:
- Multiple Myeloma Participants: Participants with MM were observed retrospectively since the diagnosis up to death or lost to follow-up within the eligibility window of time (between January 1, 2008 and December 31, 2016), in this study.
Period: Overall Study
Arm/Group | Multiple Myeloma Participants
Started | 943
Completed | 943
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants eligible for analyses were included.
Arm/Group | Multiple Myeloma Participants
Number analyzed (Participants) | 943
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 437
  Male | 506
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 576
  Race: Pardo (Mixed Race or Mulatto) | 142
  Race: Black | 63
  Race: Asian | 4
  Race: Indigenous Person | 1
  Race: Unknown | 157
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 943

OUTCOME MEASURES:

1. Primary Outcome: Number of Multiple Myeloma (MM) Participants Categorized by Clinical Characteristics
Description: MM clinical characteristics upon diagnosis were classified by eligibility criteria for transplantation (eligible/not eligible) and included: presence of plasma cells in the bone marrow by biopsy and aspiration, bone or extramedullary biopsy, plasma cells determined by immunohistochemistry (Yes/No/Unknown), plasma cells determined by flow cytometry (Yes/No/Unknown) hypercalcemia, renal failure, anemia, and bone lesions features (more than one focal lesion on magnetic resonance imaging (MRI) that is at least 5 mm or greater in size), presence of monoclonal proteins (immunoglobulin (Ig)G, IgG kappa, IgG lambda, IgA, IgA kappa, IgA lambda, kappa only, lambda only, IgD, IgE, IgM, Non-secretory and Unknown), free light chain ratio (serum involved / uninvolved free light chain ratio of 100 or greater, provided the absolute level of the involved light chain is at least 100 mg/L). Only categories with data are reported. Participants were counted multiple times in different categories.
Time Frame: From initial diagnosis up to end of follow up treatment or to the retrospective cut-off date within the time of interest (between January 1, 2008, and December 31, 2016) [approximately 11.7 years]
Population: All participants eligible for analyses were included. Number analyzed are the participants with data available for analyses of the specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma Participants
Number analyzed (Participants) | 943
Participants
  Bone Marrow Biopsy: Eligible | 342
  Bone Marrow Biopsy: Not Eligible | 366
  Bone Marrow Aspiration: Eligible | 48
  Bone Marrow Aspiration: Not Eligible | 36
  Bone or Extramedullary Biopsy: Eligible | 232
  Bone or Extramedullary Biopsy: Not Eligible | 241
  Immunohistochemistry Performed: Yes: Eligible | 161
  Immunohistochemistry Performed: Yes: Not Eligible | 142
  Immunohistochemistry Performed: No: Eligible | 245
  Immunohistochemistry Performed: No: Not Eligible | 281
  Immunohistochemistry Performed: Unknown: Eligible | 46
  Immunohistochemistry Performed: Unknown: Not Eligible | 68
  Flow Cytometry Performed: Yes: Eligible: number analyzed (Participants) | 942
  Flow Cytometry Performed: Yes: Eligible | 136
  Flow Cytometry Performed: Yes: Not Eligible: number analyzed (Participants) | 942
  Flow Cytometry Performed: Yes: Not Eligible | 130
  Flow Cytometry Performed: No: Eligible: number analyzed (Participants) | 942
  Flow Cytometry Performed: No: Eligible | 254
  Flow Cytometry Performed: No: Not Eligible: number analyzed (Participants) | 942
  Flow Cytometry Performed: No: Not Eligible | 293
  Flow Cytometry Performed: Unknown: Eligible: number analyzed (Participants) | 942
  Flow Cytometry Performed: Unknown: Eligible | 62
  Flow Cytometry Performed: Unknown: Not Eligible: number analyzed (Participants) | 942
  Flow Cytometry Performed: Unknown: Not Eligible | 67
  MM Diagnosis Definition: Bone Lesion: Eligible | 15
  MM Diagnosis Definition: Bone Lesion: Not Eligible | 35
  MM Diagnosis Definition: Anemia: Eligible | 354
  MM Diagnosis Definition: Anemia: Not Eligible | 342
  MM Diagnosis Definition: Hypercalcemia: Eligible | 286
  MM Diagnosis Definition: Hypercalcemia: Not Eligible | 343
  MM Diagnosis Definition: Renal failure: Eligible | 70
  MM Diagnosis Definition: Renal failure: Not Eligible | 74
  MM Diagnosis Definition:Serum Involved/Uninvolved Free Light Chain Ratio of >=100:Eligible | 80
  MM Diagnosis Definition:Serum Involved/Uninvolved Free Light Chain Ratio of >=100:Not Eligible | 125
  MM Diagnosis Definition: >1 Focal Lesion on MRI That is >=5mm in Size: Eligible | 4
  MM Diagnosis Definition: >1 Focal Lesion on MRI That is >=5mm in Size: Not Eligible | 17
  Monoclonal Component: IgG: Eligible | 31
  Monoclonal Component: IgG: Not Eligible | 34
  Monoclonal Component: IgG Kappa: Eligible | 138
  Monoclonal Component: IgG Kappa: Not Eligible | 152
  Monoclonal Component: IgG Lambda: Eligible | 47
  Monoclonal Component: IgG Lambda: Not Eligible | 55
  Monoclonal Component: IgA: Eligible | 18
  Monoclonal Component: IgA: Not Eligible | 17
  Monoclonal Component: IgA Kappa: Eligible | 40
  Monoclonal Component: IgA Kappa: Not Eligible | 37
  Monoclonal Component: IgA Lambda: Eligible | 32
  Monoclonal Component: IgA Lambda: Not Eligible | 24
  Monoclonal Component: Kappa Only: Eligible | 38
  Monoclonal Component: Kappa Only: Not Eligible | 42
  Monoclonal Component: Lambda Only: Eligible | 32
  Monoclonal Component: Lambda Only: Not Eligible | 22
  Monoclonal Component: IgE: Eligible | 1
  Monoclonal Component: IgE: Not Eligible | 0
  Monoclonal Component: IgM: Eligible | 2
  Monoclonal Component: IgM: Not Eligible | 2
  Monoclonal Component: Non-secretory: Eligible | 18
  Monoclonal Component: Non-secretory: Not Eligible | 10
  Monoclonal Component: Unknown: Eligible | 55
  Monoclonal Component: Unknown: Not Eligible | 96

2. Primary Outcome: Number of Multiple Myeloma (MM) Participants Categorized by Treatment Patterns
Description: Treatment patterns were collected from institutional charts [included public institution, private institution and both (90% public and 10% private) institutions] of participants in Brazil. The treatment patterns were collected as induction treatment, consolidation treatment, maintenance treatment performed at Baseline (at initial diagnosis) and as a induction treatment, maintenance treatment and type of treatment performed after transplantation, for second to tenth line of treatment. Only categories with data are reported. Participants were counted multiple times in different categories.
Time Frame: as for outcome 1
Population: All participants eligible for analyses were included. Number analyzed are the number of participants with evaluable data for given category.
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma Participants
Number analyzed (Participants) | 922
Participants
  Baseline: Induction Treatment Performed: number analyzed (Participants) | 916
  Baseline: Induction Treatment Performed: Public Institution | 394
  Baseline: Induction Treatment Performed: Private Institution | 456
  Baseline: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 66
  Baseline: Consolidation Treatment Performed: number analyzed (Participants) | 17
  Baseline: Consolidation Treatment Performed: Public Institution | 3
  Baseline: Consolidation Treatment Performed: Private Institution | 14
  Baseline: Consolidation Treatment Performed: Both (90% public and 10% private) Institutions | 0
  Baseline: Maintenance Treatment Performed: number analyzed (Participants) | 76
  Baseline: Maintenance Treatment Performed: Public Institution | 39
  Baseline: Maintenance Treatment Performed: Private Institution | 32
  Baseline: Maintenance Treatment Performed: Both (90% public and 10% private) Institutions | 5
  2nd Line: Induction Treatment Performed: number analyzed (Participants) | 495
  2nd Line: Induction Treatment Performed: Public Institution | 230
  2nd Line: Induction Treatment Performed: Private Institution | 236
  2nd Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 29
  2nd Line: Maintenance Treatment Performed: number analyzed (Participants) | 35
  2nd Line: Maintenance Treatment Performed: Public Institution | 22
  2nd Line: Maintenance Treatment Performed: Private Institution | 9
  2nd Line: Maintenance Treatment Performed: Both (90% public and 10% private) Institutions | 4
  2nd Line: Type of Treatment Performed After Transplantation: number analyzed (Participants) | 14
  2nd Line: Type of Treatment Performed After Transplantation: Public Institution | 7
  2nd Line: Type of Treatment Performed After Transplantation: Private Institution | 6
  2nd Line: Type of Treatment Performed After Transplantation: Both (90% public and 10% private) Institutions | 1
  3rd Line: Induction Treatment Performed: number analyzed (Participants) | 284
  3rd Line: Induction Treatment Performed: Public Institution | 142
  3rd Line: Induction Treatment Performed: Private Institution | 131
  3rd Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 11
  3rd Line: Maintenance Treatment Performed: number analyzed (Participants) | 18
  3rd Line: Maintenance Treatment Performed: Public Institution | 13
  3rd Line: Maintenance Treatment Performed: Private Institution | 3
  3rd Line: Maintenance Treatment Performed: Both (90% public and 10% private) Institutions | 2
  3rd Line: Type of Treatment Performed After Transplantation: number analyzed (Participants) | 3
  3rd Line: Type of Treatment Performed After Transplantation: Public Institution | 2
  3rd Line: Type of Treatment Performed After Transplantation: Private Institution | 1
  3rd Line: Type of Treatment Performed After Transplantation: Both (90% public and 10% private) Institutions | 0
  4th Line: Induction Treatment Performed: number analyzed (Participants) | 146
  4th Line: Induction Treatment Performed: Public Institution | 70
  4th Line: Induction Treatment Performed: Private Institution | 70
  4th Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 6
  4th Line: Maintenance Treatment Performed: number analyzed (Participants) | 6
  4th Line: Maintenance Treatment Performed: Public Institution | 3
  4th Line: Maintenance Treatment Performed: Private Institution | 2
  4th Line: Maintenance Treatment Performed: Both (90% public and 10% private) Institutions | 1
  4th Line: Type of Treatment Performed After Transplantation: number analyzed (Participants) | 1
  4th Line: Type of Treatment Performed After Transplantation: Public Institution | 0
  4th Line: Type of Treatment Performed After Transplantation: Private Institution | 1
  4th Line: Type of Treatment Performed After Transplantation: Both (90% public and 10% private) Institutions | 0
  5th Line: Induction Treatment Performed: number analyzed (Participants) | 78
  5th Line: Induction Treatment Performed: Public Institution | 38
  5th Line: Induction Treatment Performed: Private Institution | 37
  5th Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 3
  5th line: Maintenance Treatment Performed: number analyzed (Participants) | 3
  5th line: Maintenance Treatment Performed: Public Institution | 1
  5th line: Maintenance Treatment Performed: Private Institution | 2
  5th line: Maintenance Treatment Performed: Both (90% public and 10% private) Institutions | 0
  5th Line: Type of Treatment Performed After Transplantation: number analyzed (Participants) | 1
  5th Line: Type of Treatment Performed After Transplantation: Public Institution | 0
  5th Line: Type of Treatment Performed After Transplantation: Private Institution | 1
  5th Line: Type of Treatment Performed After Transplantation: Both (90% public and 10% private) Institutions | 0
  6th Line: Induction Treatment Performed: number analyzed (Participants) | 41
  6th Line: Induction Treatment Performed: Public Institution | 21
  6th Line: Induction Treatment Performed: Private Institution | 19
  6th Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 1
  6th Line: Maintenance Treatment Performed: number analyzed (Participants) | 2
  6th Line: Maintenance Treatment Performed: Public Institution | 2
  6th Line: Maintenance Treatment Performed: Private Institution | 0
  6th Line: Maintenance Treatment Performed: Both (90% public and 10% private) Institutions | 0
  7th Line: Induction Treatment Performed: number analyzed (Participants) | 16
  7th Line: Induction Treatment Performed: Public Institution | 6
  7th Line: Induction Treatment Performed: Private Institution | 10
  7th Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 0
  8th Line: Induction Treatment Performed: number analyzed (Participants) | 5
  8th Line: Induction Treatment Performed: Public Institution | 3
  8th Line: Induction Treatment Performed: Private Institution | 2
  8th Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 0
  9th Line: Induction Treatment Performed: number analyzed (Participants) | 3
  9th Line: Induction Treatment Performed: Public Institution | 1
  9th Line: Induction Treatment Performed: Private Institution | 2
  9th Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 0
  10th Line: Induction Treatment Performed: number analyzed (Participants) | 2
  10th Line: Induction Treatment Performed: Public Institution | 1
  10th Line: Induction Treatment Performed: Private Institution | 1
  10th Line: Induction Treatment Performed: Both (90% public and 10% private) Institutions | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time elapsed between the date of diagnosis until death, with censoring of participants who were alive when last seen or who lost to follow up.
Time Frame: From the date of diagnosis up to death within the period of interest (between January 1, 2008, and December 31, 2016) or up to the end of this study [up to 11.7 years]
Population: All participants eligible for analyses who had non-missing observations were analyzed. Number analyzed is the number of participants with data available for given category.
Measure: Median (Full Range); unit: days
Arm/Group | Multiple Myeloma Participants
Number analyzed (Participants) | 922
days
  Eligible for Transplantation but not Performed: number analyzed (Participants) | 174
  Eligible for Transplantation but not Performed | 1926 [1516 to 2834]
  Eligible for Transplantation and Performed: number analyzed (Participants) | 264
  Eligible for Transplantation and Performed | 3277 [2859 to NA] — The upper limit of 95% confidence interval were not estimable due to low number of participants with data.
  Not Eligible for Transplantation: number analyzed (Participants) | 484
  Not Eligible for Transplantation | 1566 [1367 to 1894]
Statistical Analysis 1: Comparison: Multiple Myeloma Participants; Test type: Other; p < 0.0001, Log Rank — Statistical differences among eligible performed, eligible not performed and not eligible participants were estimated by Log Rank test

4. Secondary Outcome: Duration of Treatment
Description: Duration of treatment was defined with respect to selected lines or regimens of interest, considering the time elapsed from each treatment initiation to discontinuation, and censoring participants who lost to follow-up before discontinuation. Duration of treatment was classified by participants eligibility- eligible/not eligible for transplantation. The deaths occurred after treatment initiation to end of study are reported in categories 'Since Diagnosis to Death-Eligible and Not Eligible'.
Time Frame: From treatment initiation up to discontinuation of treatment or lost to follow-up, whichever occurs first up to the end of this study (up to 11.7 years)
Population: as for outcome 3
Measure: Median (Full Range); unit: years
Arm/Group | Multiple Myeloma Participants
Number analyzed (Participants) | 922
years
  Since Diagnosis for Living Participants: Eligible: number analyzed (Participants) | 230
  Since Diagnosis for Living Participants: Eligible | 5 [0.6 to 11.7]
  Since Diagnosis for Living Participants: Not Eligible: number analyzed (Participants) | 160
  Since Diagnosis for Living Participants: Not Eligible | 4.2 [0 to 11.2]
  Since Diagnosis to Lost to Follow-up: Eligible: number analyzed (Participants) | 39
  Since Diagnosis to Lost to Follow-up: Eligible | 3.6 [0 to 8.5]
  Since Diagnosis to Lost to Follow-up: Not Eligible: number analyzed (Participants) | 68
  Since Diagnosis to Lost to Follow-up: Not Eligible | 2.3 [0.1 to 8.6]
  Since Diagnosis to Death: Eligible: number analyzed (Participants) | 169
  Since Diagnosis to Death: Eligible | 2.8 [0 to 9.9]
  Since Diagnosis to Death: Not Eligible: number analyzed (Participants) | 256
  Since Diagnosis to Death: Not Eligible | 1.8 [0 to 10]

ADVERSE EVENTS:
Time Frame: From diagnosis up to the end of this study (up to 11.7 years)
Description: Only deaths were collected, and data of adverse events or adverse drug reactions were not collected as part of the study database.
Arm/Group | Multiple Myeloma Participants
All-Cause Mortality (participants affected / at risk) | 436/943
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03506386/Prot_SAP_000.pdf